CLINICAL TRIAL: NCT03321487
Title: Safety and Feasibility of Primary Motor Cortex Blood-Brain Barrier Opening Using Transcranial MR-Guided Focused Ultrasound With Intravenous Ultrasound Contrast Agent in Patients With Amyotrophic Lateral Sclerosis
Brief Title: Blood-Brain Barrier Opening Using MR-Guided Focused Ultrasound in Patients With Amyotrophic Lateral Sclerosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: InSightec (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ALSFUS001
Record Dates: First submitted 2017-10-23; First posted 2017-10-25 (Actual); Last update posted 2021-09-08 (Actual); Status verified 2021-01

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: Blood-Brain Barrier disruption; Blood-Brain Barrier opening; magnetic resonance-guided focused ultrasound
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stage I Cohort (Experimental): Blood-Brain Barrier opening with MRgFUS. BBB opening of a small volume of the primary motor cortex
  Interventions: Device: Blood-Brain Barrier opening with MRgFUS
- Stage II Cohort (Experimental): Blood-Brain Barrier opening with MRgFUS. BBB opening of a larger volume of the primary motor cortex
  Interventions: Device: Blood-Brain Barrier opening with MRgFUS

INTERVENTIONS:
Device: Blood-Brain Barrier opening with MRgFUS — ExAblate Transcranial MR-guided Focused Ultrasound to temporarily open the Blood-Brain Barrier
  Other Names: Focused Ultrasound (FUS); Blood-Brain Barrier Disruption (BBBD); ExAblate MRgFUS

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, and feasibility of Blood-Brain Barrier (BBB) opening using transcranial MRI-guided focused ultrasound in conjunction with an intravenous ultrasound contrast agent in patients with Amyotrophic Lateral Sclerosis (ALS).

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed with laboratory supported probable, clinically probable or definite ALS according to the World Federation of Neurology Revised El Escorial criteria (Brooks et al. 2000).
2. Right-hand dominant male or female aged 18 years or older.
3. Capable of providing informed consent and complying with study procedures, including tolerability in the supine position and MRI examination without significant claustrophobia.
4. If taking riluzole, on a stable dose for at least 30 days prior to Screening Visit.
5. Slow Vital Capacity equal to or more than 50% predicted value for gender, height and age in the 30 days prior to the Screening Visit and able to lie supine without BiPAP.
6. Severe left arm weakness and functional impairment, defined as Medical Research Council muscle strength score equals 3 or less in the index finger abduction and thumb abduction on the left side; OR severe left leg weakness and functional impairment, defined as Medical Research Council muscle strength score equals 3 or less at the hip flexors and ankle dorsiflexors on the left side.
7. Able to communicate during the ExAblate® MRI-guided FUS procedure.

Exclusion Criteria:

1. Unable to complete high-density CT and MRI studies of the head at the Screening Visit or any other MRI contraindication, such as:

   * Large body habitus and not fitting comfortably into the scanner
   * Difficulty lying supine and still for up to 3 hours in the MRI unit or significant claustrophobia
2. MRI findings:

   * Active infection/inflammation
   * Acute or chronic brain hemorrhages, specifically lobar or subcortical microbleeds, siderosis or macrohemorrhages
   * Tumor/space occupying lesion
   * Meningeal enhancement
3. More than 30% of the skull area traversed by the sonication pathway is covered by scars, scalp disorders (e.g., eczema), or atrophy of the scalp.
4. Clips or other metallic implanted objects in the skull or the brain, except shunts.
5. Significant cardiac disease or unstable hemodynamic status including:

   * Documented myocardial infarction within six months of enrollment
   * Unstable angina on medication
   * Unstable or worsening congestive heart failure
   * Left ventricular ejection fraction below the lower limit of normal
   * History of a hemodynamically unstable cardiac arrhythmia
   * Cardiac or phrenic pacemaker
   * Known right-to-left, bidirectional, or transient right-to-left cardiac shunt
   * Patients with relative contraindications to perflutren including subjects with a family or personal history of QT prolongation or taking concomitant medications known to cause QTc prolongation,
   * QT prolongation observed on screening ECG (QTc > 450 for men and >470 for women)
6. Uncontrolled hypertension (systolic > 150 or diastolic BP > 100 on medication).
7. On medications that increase the bleeding risk, specifically: a) aspirin or another antiplatelet medication (clopidogrel, prasugrel, ticlopidine, abciximab) for the last 7 days prior to treatment; b) oral, subcutaneous or intravenous anticoagulant medications, such as oral vitamin K inhibitors for the last 7 days, non-vitamin K inhibitor oral anticoagulant (dabigatran, apixaban, rivaroxaban) for the last 72 hours, and intravenous or subcutaneous heparin-derived compounds for the last 48 hours.
8. History of a bleeding disorder, coagulopathy or a history of spontaneous hemorrhage.
9. Known frontotemporal dementia.
10. Abnormal coagulation profile, specifically: platelet <100,000/μl, Prothrombin Time >14 seconds, activated partial thromboplastin time (aPTT) >36 seconds, and INR > 1.3.
11. Known cerebral or systemic vasculopathy, specifically cerebral amyloid angiopathy or systemic or central nervous system vasculitis.
12. Known auto-immune condition with or without neurological manifestations (e.g., multiple sclerosis (MS), systemic lupus erythematous (SLE), Rheumatoid arthritis).
13. Current or planned use of oral, intramuscular or intravenous steroid drugs (such as prednisone, prednisolone, dexamethasone, triamcinolone, methylprednisolone, oxandrolone, and others) or immunosuppressant drugs (azathioprine, mycophenolate, tacrolimus, sirolimus, cyclophosphamide, and others) for more than 7 days.
14. Known sensitivity/allergy to gadolinium (an alternative product may be used), DEFINITY® contrast or any of its components.
15. Untreated, uncontrolled sleep apnea.
16. Impaired renal function with cystatin C-based estimated glomerular filtration rate <30 mL/min/1.73m2 and acute renal injury.
17. Currently in a clinical trial involving an investigational product or non-approved use of a drug or device.
18. Known respiratory diseases, specifically: chronic pulmonary disorders e.g., severe/uncontrolled COPD, pulmonary vasculitis, or other causes of reduced pulmonary vascular cross-sectional area, asthma or hay fever.
19. Patients with a history of drug allergies or multiple allergies where the benefit/risk of administering DEFINITY® is considered unfavorable by the study physicians in relation to the product monograph for DEFINITY®.
20. Unqualified fit for the anesthesia by an anesthesiologist assessment, ASA I-III.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Estimated)
Dates: Start 2018-04-13 (Actual); Primary Completion 2021-12-30 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
Safety - Device and Procedure related adverse events | At the time of the ExAblate MRgFUS procedure
  The number and severity of device and BBB opening procedure related adverse events will be evaluated.

SECONDARY OUTCOMES:
Degree of contrast enhancement seen on post-procedure MRI | At the time of the ExAblate MRgFUS procedure and 24 hours post-procedure
  The extent and reversibility of BBB opening will be determined by the degree of contrast enhancement seen on post-procedure MRI with gadolinium-based contrast agent.

CONTACTS AND LOCATIONS:
Overall Officials: Lorne Zinman, MD, Principal Investigator — Medical Director, ALS/Neuromuscular Clinic, Sunnybrook Health Sciences Centre
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No